CLINICAL TRIAL: NCT03850015
Title: High Frame Rate Contrast Enhanced-ultrasound for the Assessment of Ischaemic Heart Disease
Brief Title: High Frame Rate Ultrasound in Heart Disease Assessment
Acronym: RUFUS-Heart
Status: Recruiting | Type: Observational
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CRC/2018/001
Record Dates: First submitted 2019-01-30; First posted 2019-02-21 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: echocardiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Standard echocardiography — Patients will undergo standard echocardiography, with and without contrast
Other: High frame rate echocardiography — Following standard echocardiography, the test is repeated using high frame rate ultrasound

SUMMARY:
The study will compare standard ultrasound images to high frame rate ultrasound images in patients with heart disease or with a low risk of heart disease to see if a higher frame rate of ultrasound adds to the information obtained from standard ultrasound.

DETAILED DESCRIPTION:
Following informed consent, patients recruited for the study will have an IV cannula inserted and will undergo imaging using 2 ultrasound systems. Standard clinical system (Philips IE33) will be used for 2D and CE imaging, followed by imaging using the Verasonics VantageTM research system (Verasonics Inc., Redmond, WA), using both conventional 2D and HFR modes.

Baseline unenhanced 2D and Doppler images would initially be acquired using Philips IE33 system and Verasonics VatangeTM unenhanced conventional 2D and HFR mode .

Ultrasound contrast agent (Sonovue) will be then injected via the intravenous (iv) cannula and 3 sets rest contrast images will be acquired - using the Phillips IE33, Verasonics and Verasonics VantageTM platform (conventional CE and HFR CE). Both systems will be optimised separately on each patient before and during infusion of contrast agent. When the optimal imaging and destruction parameters are set, there are not modified along the acquisition.

This is followed by dipyridamole infusion and the scans being repeated during stress - 3 sets contrast images will be acquired - using the Philips IE33 and Verasonics VantageTM platform (conventional CE and HFR CE).

ELIGIBILITY:
Inclusion criteria Either

* Ability to give informed consent
* age ≥18years and
* confirmed inducible wall motion / perfusion abnormality on previous stress echocardiogram
* known coronary artery disease - defined by presence of flow-limiting coronary stenosis(>70% diameter stenosis) on coronary angiography.

OR

• patient who has been assessed as at low risk of having coronary heart disease

Exclusion Criteria:

* Inability to undertake pharmacological stress, ie previously known intolerance to dipyridamole;
* Moderate or Severe aortic or mitral regurgitation or severe mitral stenosis;
* Significant pulmonary disease like severe COPD or pulmonary fibrosis;
* Atrial fibrillation;
* Inability to provide informed consent;
* Pregnancy and lactation;
* Known allergy to Sonovue
* Patients with second and third degree heart block, unless they have a pacemaker fitted
* Systolic BP < 90
* Known Myasthenia Gravis
* Bronchial asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25 patients will be recruited over 12 months. 5 of these patients will be at low high of having coronary artery disease and 20 at high risk of coronary artery disease. patients will be recruited from those referred for clinical stress stress echocardiography.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Agreement between HFR ultrasound and standard ultrasound. | At 1 year
  Demonstration that there is at least 80% agreement between HFR ultrasound techniques and standard techniques. Expressed as as a percentage of the recorded images.

CONTACTS AND LOCATIONS:
Overall Officials: Roxy Senior, MD, Principal Investigator — LONDON NORTH WEST UNIVERSITY HEALTHCARE NHS TRUST
Locations (1):
- London North West University Healthcare NHS Trust, Harrow, Middx, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared